CLINICAL TRIAL: NCT06205992
Title: Three-dimensional MR Elastography and Two-dimensional MR Elastography for Assessing Cirrhosis and Portal Hypertension：A Prospective Multicenter Study
Brief Title: 3D-MRE and 2D-MRE for Assessing Cirrhosis and Portal Hypertension
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radology, Shengjing Hospital
Other Study IDs: ShengjingH2206
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis; Liver Portal Hypertension
Keywords: 3D-MRE; 2D-MRE; HVPG
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Experimental group was set to develop the novel non-invasive model for virtual HVPG using 3d-MRE
  Interventions: Device: 3D-MRE; Device: HVPG
- Control group: Control group was set to develop the novel non-invasive model for virtual HVPG using 2d-MRE
  Interventions: Device: 2D-MRE; Device: HVPG

INTERVENTIONS:
Device: 3D-MRE — All imaging studies were performed by using a 3.0-T MRI system (Signa HDx, GE Healthcare) with an eight-channel phasedarray body coil.
  Groups: Experimental group
Device: HVPG — HVPG measurements are performed by well-trained interventional radiologists in accordance with standard operating procedures
  Groups: Experimental group
Device: 2D-MRE — All imaging studies were performed by using a 3.0-T MRI system (Signa HDx, GE Healthcare) with an eight-channel phasedarray body coil.
  Groups: Control group
Device: HVPG — HVPG measurements are performed by well-trained interventional radiologists in accordance with standard operating procedures
  Groups: Control group

SUMMARY:
How to construct a novel, non-invasive, accurate, and convenient method to achieve prediction of hepatic venous pressure gradient (HVPG) is an important general problem in the management of portal hypertension in cirrhosis. We plan to compare the ability of three demensional-magnetic resonance elastography (3D-MRE) to two demensional-magnetic resonance elastography (2D-MRE) to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis.

DETAILED DESCRIPTION:
China suffers the heaviest burden of liver disease in the world. The number of chronic liver disease is more than 400 million. Either viral-related hepatitis, alcoholic hepatitis, or metabolic-related fatty hepatitis, etc. may progress to cirrhosis, which greatly threatens public health. Portal hypertension is a critical risk factor that correlates with clinical prognosis of patients with cirrhosis. According to the Consensus on clinical application of hepatic venous pressure gradient in China (2018), hepatic venous pressure gradient (HVPG) greater than 10,12,16,20 mmHg correspondingly predicts different outcomes of patients with cirrhosis portal hypertension. It is of great significance to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis. As a universal gold standard for diagnosing and monitoring portal hypertension, HVPG remains limitation for clinical application due to its invasiveness. How to construct a novel, non-invasive, accurate, and convenient method to achieve prediction of HVPG is an important general problem in the management of portal hypertension in cirrhosis. MR elastography allows for basic viscoelastic modeling of tissue, partitioning the complex shear modulus intoelastic components (eg, storage modulus) and viscous components (eg, lossmodulus and damping ratio [DR]). In previous studies, scholars have studied 2d MR elastography in cirrhosis to identify specific hepatic pathophysiologic interrelations. However, these mechanical properties of tissue measured with use of 3D MR elastography have yet to be investigated in cirrhosis to identify specific hepatic pathophysiologic interrelations. The investigators hypothesize that these mechanical properties might be valid presumptive surrogates of cirrhosis and portal hypertension, perhaps capable of supplanting liver biopsy or other invasive diagnostic interventions. This project aims to compare the ability of three demensional-magnetic resonance elastography (3D-MRE) to two demensional-magnetic resonance elastography (2D-MRE) to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years old
2. confirmed cirrhosis (laboratory, imaging and clinical symptoms)
3. with 3D-MRE and 2D-MRE within 1 month prior to HVPG measurement
4. written informed consent

Exclusion Criteria:

1. any previous liver or spleen surgery
2. liver cancer; chronic acute liver failure
3. acute portal hypertension
4. unreliable HVPG, 3D-MRE or 2D-MRE results due to technical reasons
5. with liver interventional therapy between HVPG and MRE

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Organize paticipating units to collect standard-of-care data including radiological and clinical data. Patients diagnosed with cirrhosis who received HVPG measurement, 3D-MRE and 2D-MRE should be enrolled
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the features of 3D-MRE and 2D-MRE for assessing portal hypertension in cirrhosis. | 12 months
  WIth HVPG as reference standand, the overall diagnostic perforemace (accuracy) for cirrhosis and portal hypertension of 3D-MRE and 2D-MRE was compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi Y, Qi YF, Lan GY, Wu Q, Ma B, Zhang XY, Ji RY, Ma YJ, Hong Y. Three-dimensional MR Elastography Depicts Liver Inflammation, Fibrosis, and Portal Hypertension in Chronic Hepatitis B or C. Radiology. 2021 Oct;301(1):154-162. doi: 10.1148/radiol.2021202804. Epub 2021 Aug 10. PMID 34374594
- [Background] Yu Q, Huang Y, Li X, Pavlides M, Liu D, Luo H, Ding H, An W, Liu F, Zuo C, Lu C, Tang T, Wang Y, Huang S, Liu C, Zheng T, Kang N, Liu C, Wang J, Akcalar S, Celebioglu E, Ustuner E, Bilgic S, Fang Q, Fu CC, Zhang R, Wang C, Wei J, Tian J, Ormeci N, Ellik Z, Asiller OO, Ju S, Qi X. An imaging-based artificial intelligence model for non-invasive grading of hepatic venous pressure gradient in cirrhotic portal hypertension. Cell Rep Med. 2022 Mar 15;3(3):100563. doi: 10.1016/j.xcrm.2022.100563. eCollection 2022 Mar 15. PMID 35492878